CLINICAL TRIAL: NCT00716859
Title: A Phase 3 Prospective, Randomized, Double-Masked, 12-Week, Parallel Group Study Evaluating The Efficacy And Safety Of Latanoprost And Timolol In Pediatric Subjects With Glaucoma.
Brief Title: A Phase 3 Prospective, Randomized, Double-Masked, 12-Week, Parallel Group Study In Pediatric Subjects With Glaucoma.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A6111137
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Results first posted 2010-12-02 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2011-01

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Timolol; Latanoprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Timolol (Active Comparator)
  Interventions: Drug: Timolol
- latanoprost (Experimental)
  Interventions: Drug: latanoprost

INTERVENTIONS:
Drug: Timolol — Timolol 0.5% dosed twice-daily
  Arms: Timolol
Drug: latanoprost — Latanoprost 0.005% ophthalmic solution dosed once-daily
  Arms: latanoprost

SUMMARY:
To assess the effectiveness of latanoprost 0.005% ophthalmic solution dosed once-daily and timolol 0.5% dosed twice-daily in paediatric subjects of 18 years of age or under who are diagnosed with glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of 18 years of age or under
* Diagnosis of glaucoma
* IOP of 22 mmHg or above in at least 1 eye

Exclusion Criteria:

* Require surgery for acute angle closure
* Have had prior cyclodestructive procedures
* Have a history of ocular trauma or surgery in either eye within 3 months of the baseline visit

Ages: 36 Weeks to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 139 (Actual)
Dates: Start 2008-07; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (43):
- United States (6):
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Henderson, Nevada
  - Pfizer Investigational Site, Las Vegas, Nevada
- Pfizer Investigational Site, Leuven, Belgium
- Colombia (2):
  - Pfizer Investigational Site, Medellín, Antioquia
  - Pfizer Investigational Site, Bogota, Cundinamarca
- Pfizer Investigational Site, Prague, Czechia
- France (3):
  - Pfizer Investigational Site, Amiens, Cedex 1
  - Pfizer Investigational Site, Lille
  - Pfizer Investigational Site, Lyon
- Germany (2):
  - Pfizer Investigational Site, Regenstauf
  - Pfizer Investigational Site, Schorndorf
- India (3):
  - Pfizer Investigational Site, Hyderabad, Andhra Pradesh
  - Pfizer Investigational Site, Ahmedabad, Gujarat
  - Pfizer Investigational Site, Coimbatore, Tamil Nadu
- Italy (2):
  - Pfizer Investigational Site, Catania
  - Pfizer Investigational Site, Milan
- Philippines (2):
  - Pfizer Investigational Site, Makati City
  - Pfizer Investigational Site, Mandaluyong
- Poland (3):
  - Pfizer Investigational Site, Bialystok
  - Pfizer Investigational Site, Gdansk
  - Pfizer Investigational Site, Wroclaw
- Portugal (3):
  - Pfizer Investigational Site, Coimbra
  - Pfizer Investigational Site, Lisbon
  - Pfizer Investigational Site, Porto
- Pfizer Investigational Site, Cluj-Napoca, Cluj, Romania
- Russia (2):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Saint Petersburg
- Pfizer Investigational Site, Belgrade, Serbia
- Pfizer Investigational Site, Bratislava, Slovakia
- Pfizer Investigational Site, Ljubljana, Slovenia
- Pfizer Investigational Site, Myfair West, South Africa
- Spain (3):
  - Pfizer Investigational Site, Esplugues de Llobregat, Barcelona
  - Pfizer Investigational Site, Madrid
  - Pfizer Investigational Site, Seville
- Ukraine (3):
  - Pfizer Investigational Site, Kharkiv
  - Pfizer Investigational Site, Kyiv
  - Pfizer Investigational Site, Odesa
- United Kingdom (2):
  - Pfizer Investigational Site, Birmingham
  - Pfizer Investigational Site, London

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6111137&StudyName=A%20Phase%203%20Prospective%2C%20Randomized%2C%20Double-Masked%2C%2012-Week%2C%20Parallel%20Group%20Study%20In%20Pediatric%20Subjects%20With%20Glaucoma.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomization was stratified by age, diagnosis (congenital glaucoma [PCG] or non-congenital glaucoma [non-PCG], and intraocular pressure [IOP]) of the study eye at baseline.
Groups:
- Timolol: Timolol maleate ophthalmic solution; 1 drop of timolol 0.5% (or optionally 0.25% for participants younger than 3 years old) at approximately 8 AM and again at approximately 8 PM .
- Latanoprost: Latanoprost ophthalmic solution and vehicle; 1 drop of vehicle daily at approximately 8 AM and 1 drop (latanoprost 0.005%) daily at approximately 8 PM.
Period: Overall Study
Arm/Group | Timolol | Latanoprost
Started | 70 | 69
Received Treatment | 69 | 68
Completed | 61 | 64
Not Completed | 9 | 5
Not completed — Adverse Event | 4 | 1
Not completed — Lack of Efficacy | 3 | 0
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Not treated | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Timolol | Latanoprost | Total
Number analyzed (Participants) | 69 | 68 | 137
Age, Customized [Number; unit: Participants]
  12 to 18 years | 23 | 25 | 48
  3 to less than (<) 12 years | 29 | 26 | 55
  0 to < 3 years | 17 | 17 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 34 | 71
  Male | 32 | 34 | 66

OUTCOME MEASURES:

1. Primary Outcome: Reduction From Baseline in Mean IOP at Week 12, Last Observation Carried Forward (LOCF)
Description: Calculated as Baseline IOP minus Week 12 IOP, LOCF. IOP measured using 1 of 3 methods: Goldmann applanation tonometry (preferred method, if feasible), Perkins tonometry, or TonoPen. IOP was measured twice and if the measurements were less than or equal to (≤) 2 millimeters of mercury (mmHg) of each other, the mean of the 2 readings was recorded as the IOP at that time point. Otherwise, a third IOP measurement was taken and the median IOP recorded.
Time Frame: Baseline, Week 12
Population: Per Protocol (PP) Population: participants with no major protocol violations who received at least 1 week of study medication and had at least Week 1 IOP measurements. LOCF.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Timolol | Latanoprost
Number analyzed (Participants) | 54 | 53
mmHg | 5.72 (0.81) | 7.18 (0.81)
Statistical Analysis 1: Comparison: Timolol vs Latanoprost; Null hypothesis: latanoprost inferior to timolol (0.5 percent [%] optionally 0.25% for participants younger than 3 years). Power calculation: assuming common standard deviation (7 mmHg), 110 participants have 84% power to demonstrate latanoprost not inferior to timolol within 3 mmHg margin, assuming latanoprost has 1 mmHg reduction more than timolol in mean change from baseline IOP; Test type: Non-Inferiority or Equivalence — If lower limit of 95% Confidence Interval (CI) for treatment difference is above non-inferiority margin, then non-inferiority concluded. If lower limit of 95% CI for treatment difference is above non-inferiority margin and above zero, then superiority concluded. The difference and 95% CI of the difference in IOP reduction (Week 12) was computed from an analysis of covariance (ANCOVA) model with treatment and baseline diagnosis as factors and baseline IOP as covariate; Mean Difference (Net) = 1.46, 95% CI 2-sided [-0.81 to 3.74]

2. Secondary Outcome: Reduction From Baseline in Mean IOP at Week 1
Description: Calculated as Baseline IOP minus Week 1 IOP (observed). IOP measured using 1 of 3 methods: Goldmann applanation tonometry (preferred method, if feasible), Perkins tonometry, or TonoPen. IOP was measured twice and if the measurements were ≤ 2 mmHg of each other, the mean of the 2 readings was recorded as the IOP at that time point. Otherwise, a third IOP measurement was taken and the median IOP recorded.
Time Frame: Baseline, Week 1
Population: PP
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Timolol | Latanoprost
Number analyzed (Participants) | 54 | 53
mmHg | 6.02 (0.83) | 6.70 (0.84)
Statistical Analysis 1: Comparison: Timolol vs Latanoprost; Test type: Superiority or Other; Mean Difference (Net) = 0.68, 95% CI 2-sided [-1.66 to 3.02]

3. Secondary Outcome: Reduction From Baseline in Mean IOP at Week 4
Description: Calculated as Baseline IOP minus Week 4 IOP (observed). IOP measured using 1 of 3 methods: Goldmann applanation tonometry (preferred method, if feasible), Perkins tonometry, or TonoPen. IOP was measured twice and if the measurements were ≤ 2 mmHg of each other, the mean of the 2 readings was recorded as the IOP at that time point. Otherwise, a third IOP measurement was taken and the median IOP recorded.
Time Frame: Baseline, Week 4
Population: Evaluable participants in PP
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Timolol | Latanoprost
Number analyzed (Participants) | 47 | 49
mmHg | 5.37 (0.94) | 6.99 (0.92)
Statistical Analysis 1: Comparison: Timolol vs Latanoprost; Test type: Superiority or Other; Mean Difference (Net) = 1.62, 95% CI 2-sided [-1.00 to 4.25]

4. Secondary Outcome: Reduction From Baseline in Mean IOP at Week 12 (Observed)
Description: Calculated as Baseline IOP minus Week 12 IOP (observed). IOP measured using 1 of 3 methods: Goldmann applanation tonometry (preferred method, if feasible), Perkins tonometry, or TonoPen. IOP was measured twice and if the measurements were ≤ 2 mmHg of each other, the mean of the 2 readings was recorded as the IOP at that time point. Otherwise, a third IOP measurement was taken and the median IOP recorded.
Time Frame: Baseline, Week 12
Population: Evaluable participants in PP
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Timolol | Latanoprost
Number analyzed (Participants) | 43 | 46
mmHg | 6.96 (0.68) | 7.75 (0.66)
Statistical Analysis 1: Comparison: Timolol vs Latanoprost; Test type: Superiority or Other; Mean Difference (Net) = 0.4085, 95% CI 2-sided [-1.10 to 2.67]

5. Secondary Outcome: Mean IOP at Baseline
Description: IOP measured using 1 of 3 methods: Goldmann applanation tonometry (preferred method, if feasible), Perkins tonometry, or TonoPen. IOP was measured twice and if the measurements were ≤ 2 mmHg of each other, the mean of the 2 readings was recorded as the IOP at that time point. Otherwise, a third IOP measurement was taken and the median IOP recorded.
Time Frame: Baseline
Population: PP
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Timolol | Latanoprost
Number analyzed (Participants) | 54 | 53
mmHg | 27.8 (6.18) | 27.3 (5.46)

6. Secondary Outcome: Mean IOP at Week 1
Description: as for outcome 5
Time Frame: Week 1
Population: PP
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Timolol | Latanoprost
Number analyzed (Participants) | 54 | 53
mmHg | 21.7 (7.99) | 20.6 (6.38)

7. Secondary Outcome: Mean IOP at Week 4
Description: as for outcome 5
Time Frame: Week 4
Population: Evaluable participants in PP
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Timolol | Latanoprost
Number analyzed (Participants) | 47 | 49
mmHg | 21.5 (7.49) | 20.1 (6.82)

8. Secondary Outcome: Mean IOP at Week 12
Description: as for outcome 5
Time Frame: Week 12
Population: Evaluable participants in PP
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Timolol | Latanoprost
Number analyzed (Participants) | 43 | 46
mmHg | 19.8 (3.50) | 19.2 (5.87)

9. Secondary Outcome: Percentage of Participants With Greater Than or Equal to (≥) 15% IOP Reduction From Baseline at Both Weeks 4 and 12
Description: Participants with ≥15% IOP reduction from baseline at both Week 4 and Week 12. Calculated as (post baseline IOP minus baseline IOP) divided by IOP, multiplied by 100%. IOP measured using 1 of 3 methods: Goldmann applanation tonometry (preferred method, if feasible), Perkins tonometry, or TonoPen. IOP was measured twice and if the measurements were ≤ 2 mmHg of each other, the mean of the 2 readings was recorded as the IOP at that time point. Otherwise, a third IOP measurement was taken and the median IOP recorded.
Time Frame: Baseline, Week 4, and Week 12
Population: Evaluable participants in PP
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Timolol | Latanoprost
Number analyzed (Participants) | 54 | 53
Percentage of participants | 52 [38 to 66] | 60 [46 to 74]
Statistical Analysis 1: Comparison: Timolol vs Latanoprost; Test type: Superiority or Other; p = 0.3315, Cochran-Mantel-Haenszel; P-value from a Cochran-Mantel-Haenszel chi-square test stratified by baseline diagnosis (PCG vs non-PCG)

10. Secondary Outcome: Percentage of Participants Discontinuing Therapy Due to a Drug-related Adverse Experience
Description: An investigator's causality assessment was the determination of whether there existed a reasonable possibility that the investigational product caused or contributed to an adverse event (AE). If the investigator did not know whether or not investigational product caused the event, then the event was handled as "related to investigational product" for reporting purposes.
Time Frame: Baseline through Week 12
Population: Intent to treat (ITT) population: all participants who were randomized into the study and received at least 1 dose of study medication.
Measure: Number; unit: Percentage of particpants
Arm/Group | Timolol | Latanoprost
Number analyzed (Participants) | 69 | 68
Percentage of particpants | 1.4 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Timolol | Latanoprost
Serious Adverse Events (participants affected / at risk) | 7/69 | 2/68
Other Adverse Events (participants affected / at risk) | 20/69 | 12/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Timolol (N=69) | Latanoprost (N=68)
Developmental glaucoma, both eyes (Congenital, familial and genetic disorders) | 1 | 0
Angle closure glaucoma, both eyes (Eye disorders) | 1 | 0
Glaucoma, both eyes (Eye disorders) | 1 | 0
Eye haemorrhage, study eye (Eye disorders) | 1 | 0
Lens dislocation, study eye (Eye disorders) | 0 | 1
Corneal perforation, fellow eye (Eye disorders) | 1 | 0
Acute tonsillitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Trabeculectomy, both eyes (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Timolol (N=69) | Latanoprost (N=68)
Conjunctival disorder, both eyes (Eye disorders) | 2 | 0
Conjunctival hyperaemia, both eyes (Eye disorders) | 3 | 1
Conjunctival hyperaemia, study eye (Eye disorders) | 3 | 2
Visual acuity reduced, study eye (Eye disorders) | 2 | 0
Pyrexia (General disorders) | 2 | 2
Influenza (Infections and infestations) | 4 | 0
Nasopharyngitis (Infections and infestations) | 5 | 4
Rhinitis (Infections and infestations) | 1 | 2
Viral infection (Infections and infestations) | 2 | 1
Headache (Nervous system disorders) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.